CLINICAL TRIAL: NCT02459613
Title: Evaluation de la rhAnnexine V-128 radiomarquée Dans le Diagnostic de l'Endocardite Infectieuse, du Thrombus Atrial et de Leurs Complications Emboliques associées
Brief Title: Assessment of Radiolabeled rhAnnexin V-128 in Infective Endocarditis
Acronym: AnnIE
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Collaborators: Advanced Accelerator Applications (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: C13-38
Record Dates: First submitted 2015-05-13; First posted 2015-06-02 (Estimated); Last update posted 2021-08-26 (Actual); Status verified 2021-08

CONDITIONS: Endocarditis; Thrombosis
Keywords: Radionuclide imaging; Annexin
MeSH Terms: conditions — Endocarditis; Thrombosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Imaging (Experimental): 99mTc Annexin V-128 SPECT
  Interventions: Drug: 99mTc-Annexin V-128 SPECT

INTERVENTIONS:
Drug: 99mTc-Annexin V-128 SPECT

SUMMARY:
Intraluminal thrombi adherent to cardiac valves or atria share a common pathophysiology involving the aggregation of activated platelets with phosphatidylserine (PS) expression on the outer layer of the thrombus. They also share common complications, i.e. damages to the underlying myocardium and embolic risk related to thrombus fragmentation. The diagnostic work-up, currently relying on morphologic imaging alone (mainly echography), lacks sensitivity and does not allow to differentiate between active (renewal and growth activity) and quiescent (scarred) thrombus. It is therefore highly desirable to develop a new approach able to non-invasively provide insight on the biological activity of thrombi and to detect embolic events in a single exam.

Annexin V is a 36 kDa endogenous glycoprotein which binds PS with nanomolar affinity. Radiolabeled Annexin V has been shown to provide molecular imaging of PS expressed by apoptotic cells or activated platelets. The ability of the imaging agent to bind mural thrombus has been established in vivo in a murine model of abdominal aortic aneurysm and ex vivo in human. It has been also shown that radiolabeled Annexin V allowed in vivo detection of vegetations and secondary pulmonary emboli with high sensitivity in various animal models of infective endocarditis.

A radiolabeling kit of annexin V complying with GMP requirements has been developed (rhAnnexine V-128, Advanced Accelerator Applications - Atreus) and is currently available. AnniE is a single centre, proof of concept, interventional, open, non-randomized study aiming at evaluating the sensitivity of 99mTc-Annexin V-128 in the detection thrombus in comparison with reference imaging in patients presenting with either: 1/ infective endocarditis or 2/ atrial thrombus. The safety of the 99mTc-Annexin V-128 will be assessed in a first phase (10 first patients enrolled). Data in relation with safety of the imaging agent will be reviewed by an independent Data and Safety Monitoring Board (DSMB); in case of positive answer, the study will continue with a second phase. The data gathered in all patients (n=120) will be used to determine outcome measures.

ELIGIBILITY:
Inclusion Criteria:

* stable clinical status
* signed informed consent
* contraception in women of childhood potential

  * Endocarditis group:
* definite ou possible endocarditis (modified Duke criteria)

  * Atrial thrombosis group:
* presence of atrial thrombosis evidenced by transesophageal echocardiography

Exclusion Criteria:

* pregnant or lactating women
* contra-indication to both MRI and CT

  * Endocarditis group:
* history of cardiac surgery in relation with the current episode
* (effective) antibiotic regimen for more than 15 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-02-05 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Diagnostic sensitivity in infective endocarditis and atrial thrombus | up to 4 weeks

SECONDARY OUTCOMES:
Diagnostic value (sensitivity and specificity) in infective endocarditis | up to 4 weeks
Diagnostic sensitivity in atrial thrombus | up to 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Le Guludec, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Bichat Hospital, Paris, France

REFERENCES:
- [Background] Benali K, Louedec L, Azzouna RB, Merceron O, Nassar P, Al Shoukr F, Petiet A, Barbato D, Michel JB, Sarda-Mantel L, Le Guludec D, Rouzet F. Preclinical validation of 99mTc-annexin A5-128 in experimental autoimmune myocarditis and infective endocarditis: comparison with 99mTc-HYNIC-annexin A5. Mol Imaging. 2014;13. doi: 10.2310/7290.2014.00049. PMID 25431156
- [Background] Rouzet F, Dominguez Hernandez M, Hervatin F, Sarda-Mantel L, Lefort A, Duval X, Louedec L, Fantin B, Le Guludec D, Michel JB. Technetium 99m-labeled annexin V scintigraphy of platelet activation in vegetations of experimental endocarditis. Circulation. 2008 Feb 12;117(6):781-9. doi: 10.1161/CIRCULATIONAHA.107.718114. Epub 2008 Jan 28. PMID 18227388
- [Background] Duval X, Iung B, Klein I, Brochet E, Thabut G, Arnoult F, Lepage L, Laissy JP, Wolff M, Leport C; IMAGE (Resonance Magnetic Imaging at the Acute Phase of Endocarditis) Study Group. Effect of early cerebral magnetic resonance imaging on clinical decisions in infective endocarditis: a prospective study. Ann Intern Med. 2010 Apr 20;152(8):497-504, W175. doi: 10.7326/0003-4819-152-8-201004200-00006. PMID 20404380
- [Background] Sarda-Mantel L, Coutard M, Rouzet F, Raguin O, Vrigneaud JM, Hervatin F, Martet G, Touat Z, Merlet P, Le Guludec D, Michel JB. 99mTc-annexin-V functional imaging of luminal thrombus activity in abdominal aortic aneurysms. Arterioscler Thromb Vasc Biol. 2006 Sep;26(9):2153-9. doi: 10.1161/01.ATV.0000237605.25666.13. Epub 2006 Jul 20. PMID 16857952